CLINICAL TRIAL: NCT04706897
Title: Opioid Sparing Anaesthesia Via Dexmedetomidine, Ketamine and Lidocaine Infusion for Prevention of Postoperative Nausea and Vomiting in Laparoscopic Gynecological Surgery
Brief Title: Opioid Sparing Anaesthesia for Prevention of Postoperative Nausea and Vomiting in Laparoscopic Gynecological Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Ibrahim Moustafa, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 33362/9/19
Record Dates: First submitted 2021-01-10; First posted 2021-01-13 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: PONV; Opioid Sparing Anaesthesia
Keywords: Laparoscopic Gynecological Surgery; Dexmedetomidine; Ketamine; Lidocaine; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexmedetomidine; Ketamine; Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal saline (Control) group (Sham Comparator): A loading infusion of the 50 ml syringe (A) containing normal saline was started at rate of 0.2 ml/ kg/hr ten minutes before induction (as masking for mixture in group S). Then anesthesia was induced with 2 mg/kg ideal body weight (IBW) of propofol , patients were intubated with the aid of 0.5 mg/kg IBW atracurium and received 0.1ml/kg from syringe (C) containing fentanyl (1 mic/kg of IBW).
  Interventions: Drug: Normal saline
- Dexmedetomidine, ketamine and lidocaine (Study) group (Experimental): A loading infusion of syringe (B) containing the mixture was started at rate of 0.2 ml/kg/h ten minutes before induction. Then anesthesia was induced with 2 mg/kg IBW of propofol, patients were intubated with the aid of 0.5 mg/kg IBW atracurium and received 0.1ml/kg from syringe (D) containing normal saline (as masking for fentanyl in the control group).
  Interventions: Drug: Dexmedetomidine, ketamine and lidocaine

INTERVENTIONS:
Drug: Dexmedetomidine, ketamine and lidocaine — A loading infusion of syringe (B) containing the a mixture [dexmedetomidine (2 µg/ml), ketamine (0.5 mg /ml) and lidocaine (4 mg /ml)] was started at rate of 0.2 ml/kg/h ten minutes before induction. Then anesthesia was induced with 2 mg/kg IBW of propofol, patients were intubated with the aid of 0.5 mg/kg IBW atracurium and received 0.1ml/kg from syringe (D) containing normal saline (as masking for fentanyl in the control group).
  Arms: Dexmedetomidine, ketamine and lidocaine (Study) group
Drug: Normal saline — A loading infusion of the 50 ml syringe (A) containing normal saline was started at rate of 0.2 ml/ kg/hr ten minutes before induction (as masking for mixture in group S). Then anesthesia was induced with 2 mg/kg ideal body weight (IBW) of propofol , patients were intubated with the aid of 0.5 mg/kg IBW atracurium and received 0.1ml/kg from syringe (C) containing fentanyl (1mic/kg of IBW).
  Arms: Normal saline (Control) group

SUMMARY:
In spite of multimodal analgesic strategies, which consist of opioids, dexamethasone, non-steroidal anti-inflammatory drugs, and local anesthetics applied into the surgical wound, postoperative pain and postoperative nausea and vomiting (PONV) are still common complaints reported after laparoscopic gynecological surgery.

So, it is hypothesized that the infusion consisting of lidocaine, dexmedetomidine and ketamine, as an opioid substitute was a feasible technique for laparoscopic gynecological surgery and would be associated with less incidence of PONV and lower opioid requirements in the early postoperative period.

The aim of this study was to evaluate the effect of opioid sparing technique via infusion of Dexmedetomidine, Ketamine and Lidocaine on post-operative nausea and vomiting in laparoscopic gynecological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic gynaecological surgery, who:

  * had the American Society of Anesthesiologists (ASA) I or II physical status,
  * were 21-60 years of age

Exclusion Criteria:

* A body mass index >35 kg/ m2
* Pregnant, breast feeding women
* Hepatic, renal or cardiac insufficiency
* Diabetes mellitus
* History of chronic pain
* Alcohol or drug abuse
* Psychiatric disease
* Allergy or contraindication to any of the study drugs

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Laparoscopic Gynecological Surgery
Enrollment: 80 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative nausea and vomiting (PONV) | First 24 hours postoperative
  The total simplified PONV impact scale score ≥ 5

SECONDARY OUTCOMES:
Intraoperative isoflurane consumption | Intraoperative 3 hours
Intraoperative fentanyl consumption | Intraoperative 3 hours
Postoperative 24 hours morphine consumption. | First 24 hours postoperative
  First 24 hr morphine consumption according to visual analogue sale (VAS). If VAS is more than 3, Intravenous morphine titration was administered as a bolus of 2 mg (body weight ≤60 kg) or 3 mg (body weight >60 kg) with 5-minute lockout interval between each bolus repeated till pain is relieved.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta University, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP